CLINICAL TRIAL: NCT02347579
Title: Neurophysiological Basis of Rehabilitation in Complex Regional Pain Syndrome, Type I and Chronic Low Back Pain
Acronym: BrainEXPain
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: NL35546.068.11
Record Dates: First submitted 2015-01-08; First posted 2015-01-27 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with CRPS: Patients with Complex Regional Pain Syndrome, Type I
- Patients with CLBP: Patients with chronic low back pain
- Healthy controls

SUMMARY:
Complex Regional Pain syndrome Type I (CRPS-I) is a chronic progressive disease. Patients experience dramatic decline of overall well-being, despite the absence of any apparent physical cause. The main symptoms are hypersensitivity to pain (hyperalgesia) and experiencing normal tactile stimulation as painful (allodynia) in the absence of peripheral nerve damage. The debate on the aetiology of CRPS-I is still open.

The therapy offered to CRPS-I patients is diverse and can involve invasive and non-invasive interventions. Current (inter)national guidelines recommend physiotherapy as the best non-invasive treatment for rehabilitation. Recently, cognitive and behavioural Graded Exposure in Vivo (GEXP) therapy aimed at reducing pain-related fear was found to be effective (De Jong et al. 2005), and more effective than standard physical therapy (ReMOVE study, articles in preparation). By reducing pain-related fear EXP might reconcile motor output and sensory feedback.

Another type of pain is lower back pain (LBP), which affects 70% to 85% of general population, but usually heals within 12 weeks in 90% of patients. The rest of the patients suffer from intractable, chronic LBP despite no evident organic abnormality. Research shows that also in these patients cognitive and behavioural aspects of pain are important and related to physical performance and self-reported disability (Vlaeyen et al., 2000). Several studies have demonstrated the success of GEXP in this patient group: GEXP resulted in improvements in pain-related fear, catastrophizing, performance of daily relevant activities, and in pain intensity (Leeuw et al., 2008).

This study aims to investigate the effect of GEXP on brain regions involved in the processing of harmless tactile stimuli in CRPS-I and CLBP patients, as well as its effect on tactile discrimination thresholds. We hypothesize that GEXP will induce 1) an improvement of tactile discrimination thresholds, 2) a functional reorganization of primary and secondary somatosensory cortex (in regions related to the affected limb in CRPS-I; and to the back in LBP), 3) changes in activation of emotional brain circuits during non-noxious stimulation, 4) changes in resting state connectivity between emotional and sensory brain areas, 5) changes in measures reflecting white matter integrity. No systematic changes are expected in the healthy controls.

Patients diagnosed with CRPS-I and CLBP will participate in a Magnetic Resonance Imaging (MRI) experiment. In this observational study, we examine the effects of GEXP treatment that all patients receive as part of usual care. Anatomical as well as diffusion-weighted and T2*-weighted (Blood oxygenation level dependent) MR images will be acquired. The study has a 3x4 split plot design with group (CRPS-I patients and CLBP receiving GEXP treatment / healthy controls) as between-subjects variable and time (pre-, during, post-treatment and follow-up) as within-subject variable.

ELIGIBILITY:
Inclusion Criteria:

CRPS-I patients:

* A clinical diagnosis of CRPS-I according to 'the Budapest criteria' for research purposes (Harden et al., 2007):

  * Continuing pain, which is disproportionate to any inciting event
  * Must report at least one symptom in all of the four following categories:

    * Sensory: Reports of hyperesthesia and/or allodynia
    * Vasomotor: Reports of temperature asymmetry and/or skin color changes and/or skin color asymmetry
    * Sudomotor / Edema: Reports of edema and/or sweating changes and/or sweating asymmetry
    * Motor / Trophic: Reports of decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin)
  * Must display at least one sign at time of evaluation in two or more of the following categories:

    * Sensory: Evidence of hyperalgesia (to pinprick) and/or allodynia (to light touch and/or temperature sensation and/or deep somatic pressure and/or joint movement)
    * Vasomotor: Evidence of temperature asymmetry and/or skin color changes and/or asymmetry
    * Sudomotor / Edema: Evidence of edema and/or sweating changes and/or sweating asymmetry
    * Motor / Trophic: Evidence of decreased range of motion and/or motor dysfunction (weakness, tremor, dystonia) and/or trophic changes (hair, nail, skin)
  * There is no other diagnosis that better explains the signs and symptoms
* Unilateral localization on upper or lower extremity

CLBP patients:

* Experience of non-specific lower back pain for at least three months
* No other diagnosis better explaining the signs and symptoms. both patient groups:
* Report of substantial fear of movement/(re)-injury
* Age between 18 and 65 years
* Stable medication

healthy controls:

* Age between 18 and 65 years
* Matched for age, gender and handedness

Exclusion Criteria:

patients and healthy controls:

* Neuropathy of the upper or lower extremities
* MRI incompatible health condition (e. g. pacemaker, metal prosthetic devices)
* Psychiatric condition and ongoing medication that would alter emotional/sensory processing
* Previous tactile impairment in the upper or lower extremity caused by:

  * damage to the sensory apparatus
  * CNS lesion

healthy controls:

• (history of) CRPS or other chronic pain syndromes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People diagnosed with CRPS, type I, and people with chronic low back pain (CLBP) are target population for this study. A group of healthy controls matched for age, gender and handedness will also take part in the study.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline blood oxygenation level dependent (BOLD) signal (fMRI) during tactile stimulation and during rest | participants will be assessed repeatedly during the treatment; at baseline, at 5/6 weeks after start of treatment, at end of treatment (approximately 10 weeks after start) and at follow-up (6 months after end of treatment)
Change from baseline diffusion MRI measures (fractional anisotropy, neurite density, orientation dispersion) | participants will be assessed repeatedly during the treatment; at baseline, at 5/6 weeks after start of treatment, at end of treatment (approximately 10 weeks after start) and at follow-up (6 months after end of treatment)
Change from baseline tactile discrimination threshold in mm | participants will be assessed repeatedly during the treatment; at baseline, at 5/6 weeks after start of treatment, at end of treatment (approximately 10 weeks after start) and at follow-up (6 months after end of treatment)

SECONDARY OUTCOMES:
Change from baseline pain-related fear (TSK, PHODA) | participants will be assessed repeatedly during the treatment; at baseline, at 5/6 weeks after start of treatment, at end of treatment (approximately 10 weeks after start) and at follow-up (6 months after end of treatment)
Change from baseline pain catastrophizing (PCS) | participants will be assessed repeatedly during the treatment; at baseline, at 5/6 weeks after start of treatment, at end of treatment (approximately 10 weeks after start) and at follow-up (6 months after end of treatment)
Change from baseline pain intensity level as assessed on visual analog scale | daily

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands